CLINICAL TRIAL: NCT01737281
Title: Proactive Outreach for Smokers in VA Mental Health
Acronym: PROMH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIR 11-291; 1I01HX000817-01A2 (NIH)
Record Dates: First submitted 2012-11-27; First posted 2012-11-29 (Estimated); Results first posted 2019-03-14 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Smoking
Keywords: Smoking; Tobacco control; Counseling; mental health
MeSH Terms: conditions — Smoking; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Proactive outreach (Experimental): Proactive outreach to deliver 7 sessions of telephone counseling and nicotine replacement therapy.
  Interventions: Behavioral: Proactive outreach
- Usual care (Active Comparator): Usual smoking cessation care from clinical staff
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Proactive outreach — Proactive contact (mail and phone) offering smoking cessation medications and telephone counseling.
  Arms: Proactive outreach
Behavioral: Usual care — Usual smoking cessation care from VA clinical staff.
  Arms: Usual care

SUMMARY:
Veterans with a mental health diagnosis have higher a prevalence of smoking and higher rates of smoking-related morbidities compared to the general Veteran population. Smoking cessation treatment delivery in the VA typically depends on a visit from a health care provider. In this study, investigators will use information within the electronic medical record to identify all smokers with a mental health diagnosis at a VA health care facility and proactively reach out to enroll them in an intensive tobacco cessation treatment program. This approach could be generalized to other behaviors and provides a novel method to improve the health of an entire population of patients.

DETAILED DESCRIPTION:
Background:

Tobacco use is the leading preventable cause of death in the United States and contributes up to 24% of all VA healthcare costs. Veterans enrolled in the VA healthcare system smoke substantially more than the general population, which is particularly true among Veterans diagnosed with mental illness. Patients with bipolar disorder or schizophrenia have the highest smoking rates (69% and 58-90%, respectively) followed by those with PTSD (45-63%) and depression (31-51%). Numerous barriers exist for tobacco cessation among mental health patients, including high nicotine dependency, low rates of follow through for referrals, and limited availability of tobacco treatment tailored to their needs.

Rationale:

Most medical care providers assess tobacco use and advise smokers to quit, but they have insufficient time to follow up with treatment, leading to low long-term quit rates. Mental health providers who often meet regularly with patients report that they find tobacco cessation outside the scope of their practice and neither assess tobacco use nor refer smokers for treatment. These practice patterns have been very difficult to change even with intensive methods and across various settings and provider types. Therefore, the investigators here propose to use the electronic medical record system to identify smokers receiving mental health care and proactively reach out to engage them in treatment in line with the following aims:

Specific Aims:

1. Compare the reach and efficacy of a proactive outreach telephone-based tobacco cessation (PRO) program for patients seen in mental health to usual care (UC) advice and referral to local VA and community tobacco cessation resources.
2. Model longitudinal associations between baseline sociodemographic, medical and mental health characteristics and abstinence at 6 and 12 months in the PRO and UC conditions.

Methods:

Investigators will use the electronic medical record to identify N=6,400 patients across 4 VA healthcare facilities who have a clinical reminder code indicating current tobacco use in the past year and who have had a mental health visit in the past 6 months. Investigators will send each patient an introductory letter and baseline survey. Respondents will be randomized in a 1:1 fashion to intervention or control. Control participants will receive VA usual care. Intervention participants will receive proactive telephone counseling and cessation medications. Investigators will assess tobacco use at 6 and 12 months from enrollment. The primary outcome is cotinine-validated abstinence at the 12-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Current smoker (i.e., any tobacco use in past 30 days)
* Seen in VA Mental Health Clinic in prior 12 months

Exclusion Criteria:

* Dementia
* Does not speak English
* Does not have a telephone and mailing address (necessary to mail out consent materials and to deliver the telephone-based intervention)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1938 (Actual)
Dates: Start 2014-07-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2018-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott E Sherman, MD MPH, Principal Investigator — Manhattan Campus of the VA NY Harbor Healthcare System, New York, NY; Steven S. Fu, MD MSCE, Principal Investigator — Minneapolis VA Health Care System, Minneapolis, MN
Locations (4):
- United States (4):
  - James A. Haley Veterans' Hospital, Tampa, FL, Tampa, Florida
  - Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota
  - Manhattan Campus of the VA NY Harbor Healthcare System, New York, NY, New York, New York
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rogers ES, Fu SS, Krebs P, Noorbaloochi S, Nugent SM, Rao R, Schlede C, Sherman SE. Proactive outreach for smokers using VHA mental health clinics: protocol for a patient-randomized clinical trial. BMC Public Health. 2014 Dec 17;14:1294. doi: 10.1186/1471-2458-14-1294. PMID 25518878
- [Result] Hammett P, Fu SS, Lando HA, Owen G, Okuyemi KS. The association of military discharge variables with smoking status among homeless Veterans. Prev Med. 2015 Dec;81:275-80. doi: 10.1016/j.ypmed.2015.09.007. Epub 2015 Sep 21. PMID 26400636
- [Result] Rogers ES, Fu SS, Krebs P, Noorbaloochi S, Nugent SM, Gravely A, Sherman SE. Proactive Tobacco Treatment for Smokers Using Veterans Administration Mental Health Clinics. Am J Prev Med. 2018 May;54(5):620-629. doi: 10.1016/j.amepre.2018.02.011. Epub 2018 Mar 15. PMID 29551324
- [Derived] Japuntich SJ, Hammett PJ, Rogers ES, Fu S, Burgess DJ, El Shahawy O, Melzer AC, Noorbaloochi S, Krebs P, Sherman SE. Effectiveness of Proactive Tobacco Cessation Treatment Outreach Among Smokers With Serious Mental Illness. Nicotine Tob Res. 2020 Aug 24;22(9):1433-1438. doi: 10.1093/ntr/ntaa013. PMID 31957794

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Proactive Outreach | Usual Care
Started | 969 | 969
Completed | 603 | 689
Not Completed | 366 | 280

BASELINE CHARACTERISTICS:
Groups:
- Proactive Outreach: Intervention arm participants received: (1) 12 sessions of proactive telephone cessation counseling, (2) coordination of cessation medications from a VA provider, (3) mailed stress reduction materials, (4) engagement of their regular mental health provider in the treatment process through CPRS progress notes, to which their provider will be added as signer.
- Usual Care: Control arm participants received a mailed list of local VA and non-VA smoking cessation services that they can access on their own. In addition, patients randomized to the control group received treatment or referrals to treatment from their regular VA providers as part of usual care. Pharmacotherapy is available at all sites in the form of nicotine replacement (patches, gum and lozenges) and bupropion.
- Total: Total of all reporting groups
Arm/Group | Proactive Outreach | Usual Care | Total
Number analyzed (Participants) | 969 | 969 | 1938
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 662 | 646 | 1308
  >=65 years | 307 | 323 | 630
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (11.6) | 58.9 (11.3) | 58.6 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 128 | 125 | 253
  Male | 841 | 844 | 1685
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 7 | 6 | 13
  Asian | 6 | 8 | 14
  Native Hawaiian or Other Pacific Islander | 4 | 5 | 9
  Black or African American | 294 | 309 | 603
  White | 603 | 595 | 1198
  More than one race | 44 | 35 | 79
  Unknown or Not Reported | 11 | 11 | 22
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 969 | 969 | 1938

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Cotinine-Validated Abstinence From Smoking
Description: The primary outcome will be cotinine-validated abstinence from smoking at 12-month follow-up.
Time Frame: 12 months
Population: Cotinine samples were obtained by mail from 53/76 people reporting abstinence in the intervention arm and 44/58 people reporting abstinence in the control arm. Note that this reflects a "complete case analysis", only including people for whom outcome data are available.
Measure: Count of Participants; unit: Participants
Arm/Group | Proactive Outreach | Usual Care
Number analyzed (Participants) | 53 | 44
Participants | 36 | 30

2. Secondary Outcome: Number of Participants Self-Reporting 7-Day Abstinence From Cigarettes
Description: At 12 month follow-up, participants were asked if the had smoked any cigarettes in the last 7 days
Time Frame: 12 months
Population: We used a "complete case" analysis, excluding participants for whom information was not available at 12 month follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Proactive Outreach | Usual Care
Number analyzed (Participants) | 620 | 701
Participants | 119 | 96

ADVERSE EVENTS:
Time Frame: Total adverse events were based on the results form 12 month follow-up
Description: Standard adverse even definitions were used
Groups:
- Intervention Arm: Intervention arm participants received: (1) 12 sessions of proactive telephone cessation counseling, (2) coordination of cessation medications from a VA provider, (3) mailed stress reduction materials, (4) engagement of their regular mental health provider in the treatment process through CPRS progress notes, to which their provider will be added as signer.
- Control Arm: Control arm participants received a mailed list of local VA and non-VA smoking cessation services that they can access on their own. In addition, patients randomized to the control group received treatment or referrals to treatment from their regular VA providers as part of usual care. Pharmacotherapy is available at all sites in the form of nicotine replacement (patches, gum and lozenges) and bupropion.
Arm/Group | Intervention Arm | Control Arm
All-Cause Mortality (participants affected / at risk) | 9/969 | 12/969
Serious Adverse Events (participants affected / at risk) | 39/969 | 28/969
Other Adverse Events (participants affected / at risk) | 0/969 | 0/969
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention Arm (N=969) | Control Arm (N=969)
Hospitalization (Surgical and medical procedures) | 39 | 27
Life-threating event (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-08): https://cdn.clinicaltrials.gov/large-docs/81/NCT01737281/Prot_SAP_000.pdf